CLINICAL TRIAL: NCT02094651
Title: Treatment of Children With Autism Spectrum Disorders and Epileptiform EEG With Divalproex Sodium
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No eligible patients were enrolled
Sponsor: Boston Children's Hospital (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Principal Investigator, Sarah Spence, Assistant in Neurology, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P00005744
Record Dates: First submitted 2014-03-10; First posted 2014-03-24 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Autism
Keywords: Abnormal EEGs
MeSH Terms: conditions — Autistic Disorder | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- divalproex sodium (Experimental): divalproex sodium will be administered in sprinkle capsule formulation, target dose of 30mg/kg, drug will be administered for 12 weeks
  Interventions: Drug: divalproex sodium
- Placebo (Placebo Comparator): Blue and white capsules with equivalent amount of lactose spheres/beads inside Placebo will be formulated to look identical to the active medication
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: divalproex sodium — The drug is an FDA approved medication for seizures but has not been approved for the treatment of epileptiform EEG abnormalities in the absence of clinical seizures.
  Other Names: Depakote; valproic acid; VPA; sodium valproate
  Arms: divalproex sodium
Other: Placebo — The placebo is an inactive substance that looks like the active drug.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if treatment of epileptiform abnormalities in children with autism spectrum disorder will improve any behaviors in these children. The investigators will study a number of different behavioral outcomes including behaviors related to attention, social communication, repetitive behaviors, maladaptive behaviors, language, motor and sensory, and sleep. The investigators will use an anticonvulsant medication called valproic acid (in the form of sodium divalproex).

DETAILED DESCRIPTION:
Epilepsy and epileptiform EEG abnormalities are common co-morbidities in Autism Spectrum Disorders (ASD) that can be considered important biomarkers of cortical dysfunction in these disorders. They may represent a measure of the excitatory-inhibitory imbalance posited to be involved in the pathogenesis of the disorder. Treatment of epilepsy is always indicated, but treatment of isolated epileptiform EEG (i.e. in the absence of clinical seizures) is frankly controversial. Since data suggest that these epileptiform discharges are associated with deficits in attention, language and behavior, the investigators believe that they may represent an important and novel treatment target in this population. The proposed study brings together a group of investigators long interested in this problem in order to investigate the efficacy of using an anticonvulsant medication with spike suppression capabilities (VPA in the form of divalproex sodium) to treat children with ASD and isolated epileptiform EEGs. Recruiting from 3 large autism centers (Boston Children's Hospital (BCH) and Vanderbilt University (VU) and University of Louisville (U of L)) with very large pediatric epilepsy units, the investigators propose a 26 week randomized placebo controlled cross over study of VPA in 4-8 year old children with ASD with frequent epileptiform EEG discharges.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 4 to 10 years.
2. Diagnosis of with ASD (Autistic Disorder, Asperger's Disorder, or pervasive developmental disorder (PDD-NOS).
3. Frequent epileptiform discharges on EEG (defined as spikes, spike wave, and sharp waves occurring at greater than 15 events per hour).
4. Intelligence quotient (IQ) range 40 to 100.
5. Weight > or = 12.5 kg.
6. English speaking families

Exclusion Criteria:

1. History of epilepsy, known neurogenetic disorder or chromosomal abnormalities with high rates of epilepsy (15q duplication syndrome, 16p deletion/duplication syndrome, Fragile X, tuberous sclerosis complex), or structural brain lesion (prior stroke, migrational defects, brain malformations).
2. The presence of a severe epileptiform EEG on the sleep EEG referred to as electrical status epilepticus in sleep (ESES) in sleep
3. Previous treatment with divalproex sodium that is any one of the following:

   * of greater than 6 months duration
   * within the last 12 months
   * that was associated with significant side effects leading to termination of treatment
4. Children who have had general anesthesia within the six months or sedation within 2 weeks of study enrollment.
5. Recent (less than two months prior to study entry) initiation of a behavioral therapy program or new psychotropic medication, or the plan to change or start a new therapy.
6. Presence of medical condition, such as carnitine deficiency, urea cycle disorder or other metabolic disorder that would be a contraindication to divalproex sodium usage.
7. Presence of a significant untreated medical problem (obstructive sleep apnea, restless legs syndrome, GERD, etc.) which may have significant impact on sleep study measures.
8. Renal, hepatic, pancreatic, or hematologic dysfunction as evidenced by values above upper limits of normal for BUN/creatinine, or values twice the upper limit of normal for serum transaminases (ALT/SGPT, AST/SGOT), values twice the upper limit of normal for serum lipase and amylase, platelets <80,000 /mcL, WBC<3.0 103 /mcL.
9. Concomitant use of medication contraindicated with divalproex sodium including topiramate, lamotrigine, and drugs that inhibit cytochrome p450 enzymes.
10. Behavioral management issues (e.g. self-injury, aggressiveness) severe enough to be of safety concerns (to subject and/or staff).
11. Absence of primary care physician.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
effect of drug vs placebo on reduction in epileptiform EEG discharges in children with ASD | In this crossover study participants will be on drug and placebo for 12 weeks each
  To examine the effect of divalproex sodium (valproate or VPA) on epileptiform EEG discharges in children with ASD. The investigators hypothesize that VPA will significantly reduce discharge counts (primary outcome measure) compared to placebo.

SECONDARY OUTCOMES:
behavior changes in drug vs placebo. | In this crossover study participants will be on drug and placebo for 12 weeks each
  To determine if administration of VPA results in improvement in behavior compared to placebo. Based on preliminary data the investigators hypothesize that VPA will be significantly associated with improvement in the areas of aggression, attention and externalizing behaviors as measured by the Child Behavior Checklist (CBCL), the primary behavioral outcome variables. A wide range of other behavioral measures (secondary outcomes) including those related to core ASD symptoms, language, adaptive functioning, sensory and motor behaviors to identify will also be examined. Behavioral measures will be examined in relation to reduction of epileptiform discharges. The investigators will also include both objective and subjective measures of sleep and examine the effect of sleep changes in relation to EEG discharge profiles and behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Spence, MD PhD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - University of Louisville, Louisville, Kentucky
  - Boston Childrens Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No